CLINICAL TRIAL: NCT02095548
Title: A Phase 1, Placebo-Controlled, Double-Blind, Dose-Escalation Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SM04690 Injected in the Target Knee Joint of Moderately to Severely Symptomatic Osteoarthritis Subjects
Brief Title: Phase 1, Dose Escalation Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SM04690 in Moderate to Severe Knee Osteoarthritis (OA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SM04690-01
Record Dates: First submitted 2014-03-18; First posted 2014-03-26 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Moderate to Severe Osteoarthritis
MeSH Terms: interventions — lorecivivint

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- SM04690, 0.03mg/2mL (Experimental): Single, intra-articular injection of SM04690, 0.03mg/2mL
  Interventions: Drug: SM04690, 0.03mg/2mL
- SM04690, 0.07mg/2mL (Experimental): Single, intra-articular injection of SM04690, 0.07mg/2mL
  Interventions: Drug: SM04690, 0.07mg/2mL
- SM04690, 0.23mg/2mL (Experimental): Single, intra-articular injection of SM04690, 0.23mg/2mL
  Interventions: Drug: SM04690, 0.23mg/2mL
- Placebo (Placebo Comparator): Single, intra-articular injection of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SM04690, 0.03mg/2mL
  Arms: SM04690, 0.03mg/2mL
Drug: SM04690, 0.07mg/2mL
  Arms: SM04690, 0.07mg/2mL
Drug: SM04690, 0.23mg/2mL
  Arms: SM04690, 0.23mg/2mL
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to find the optimal dose of SM04690 that can be safely given by intra-articular injection into the target knee joint of subjects with moderate to severe osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary OA in target knee by American College of Rheumatology (ACR) criteria
* Screening pain criteria sufficient as assessed by WOMAC and VAS scores
* Ability to read and understand the informed consent

Exclusion Criteria:

* Women who are pregnant or lactating or child bearing potential, men must use a barrier method of contraception
* Any condition, including laboratory findings, that in the opinion of the investigator constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct or evaluation
* Body mass index >40
* Major knee surgery in the target knee within 12 months prior to study or planned surgery during the study period
* History of malignancy within the last 5 years
* Participation in a clinical research trial within 12 weeks prior
* Treatment of the target knee with intra-articular steroids within 2 months or hyaluronic acid derivatives within 6 months
* Effusion of the target knee requiring aspiration within 3 months
* Use of electrotherapy or acupuncture for OA within 4 weeks
* Significant and clinically evident misalignment of the target knee
* Any known active infections
* Any chronic condition that has not been well controlled for a minimum of 3 months

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety assessments for this study will include adverse events, dose limiting toxicity (DLT), physical exams, vital signs, ECGs, and clinical laboratory tests | during 24 weeks
Additional safety assessment of bone loss as measured by CT of the knee | during 24 weeks
The following PK parameters will be determined from the plasma of SM04690; Cmax, Tmax, AUC0-t, AUC0-∞, and t1/2 | during 12 weeks

SECONDARY OUTCOMES:
Change from baseline pain over the last 48 hours using a Visual Analog Scale (VAS) | during 24 weeks
Change from baseline per Western Ontario and McMaster Osteoarthritis (WOMAC) assessment of disease scale | During 24 weeks
Change from baseline per physician global assessment of disease scale | during 24 weeks
Change from baseline in joint space width as measured by X-ray | during 24 weeks
Change from baseline of cartilage volume and thickness as measure by MRI | during 24 weeks
Change from baseline of biomarkers of cartilage synthesis and cytokines | during 24 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Tucson, Arizona
  - El Cajon, California
  - Walnut Creek, California
  - Miami, Florida
  - Boston, Massachusetts
  - Duncansville, Pennsylvania
  - Dallas, Texas

REFERENCES:
- [Derived] Yazici Y, McAlindon TE, Fleischmann R, Gibofsky A, Lane NE, Kivitz AJ, Skrepnik N, Armas E, Swearingen CJ, DiFrancesco A, Tambiah JRS, Hood J, Hochberg MC. A novel Wnt pathway inhibitor, SM04690, for the treatment of moderate to severe osteoarthritis of the knee: results of a 24-week, randomized, controlled, phase 1 study. Osteoarthritis Cartilage. 2017 Oct;25(10):1598-1606. doi: 10.1016/j.joca.2017.07.006. Epub 2017 Jul 13. PMID 28711582